CLINICAL TRIAL: NCT02319421
Title: Reducine the Risk of Alarm Fatigue Through the Use of Focused Management in Safety Huddles
Brief Title: Reducing the Risk of Alarm Fatigue Through the Use of Focused Management in Safety Huddles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-010928
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Clinical Alarms
Keywords: Alarm fatigue
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary Subjects (Experimental): Physicians and nurse practitioners caring for patients in the Pediatric Intensive Care Unit (PICU). An alarm reduction script will be used to help facilitate discussion of alarm data during weekday morning team "huddles".
  Interventions: Other: Alarm Reduction Script

INTERVENTIONS:
Other: Alarm Reduction Script — The intervention will consist of a script to facilitate the discussion of the alarm data that will take place on weekday mornings. The script will be used by huddle participants as a structured outline to rapidly discuss the high alarm low acuity patients eligible for intervention. The patients who are identified will have further discussion on rounds to determine if there are appropriate ways to reduce the alarm rates of individual patients through the safe adjustment of physiologic monitor parameters.

SUMMARY:
Context: Alarm fatigue is a threat to hospital patient safety. National surveys reveal that high alarm rates interrupt patient care, reduce trust in alarms, and lead clinicians to disable alarms entirely. Safety huddles offer an appropriate forum for reviewing alarm data and identifying patients whose high alarm rates may necessitate safe tailoring of alarm limits.

Objectives: To evaluate the impact of a focused physiologic monitor alarm reduction intervention integrated into safety huddles that involves discussing safe monitor parameter adjustments on the physiologic monitor alarm rates of individual patients with high alarm rates who meet "low acuity" criteria.

Study Design: A prospective, quasi-experimental pilot study of the impact of the huddle intervention on the alarm rates of low acuity high alarm rate individual patients discussed in huddles in the PICU. The huddle intervention will consist of a script to facilitate the discussion of the alarm data.

Setting/Participants: Participants will include all low acuity patients and their providers in the PICU at The Children's Hospital of Philadelphia.

Study Interventions and Measures: The primary outcome is the rate of crisis and warning alarms per patient day for intervention cases as compared with others in the high alarm / low acuity cohort. Safety measures will include unexpected changes in patient acuity or code blue events within one week of monitor change or discharge.

ELIGIBILITY:
Eligible primary participants will be the physicians and nurse practitioners caring for the PICU patients who are discussed as part of the huddle interventions. Eligible secondary participants will include all low acuity patients in the PICU at The Children's Hospital of Philadelphia.

Inclusion Criteria Primary Subjects: Any physician or nurse practioner caring for an intervention patient or control patient in the PICU at CHOP

Secondary Subjects:

* Low acuity patients as determined by Optilink Guidelines
* High alarm patients (top 10-20%)
* Admission to the PICU

Exclusion Criteria Primary Subjects: None

Secondary Subjects: Patients who are medically ready for transfer out of ICU or discharge home (status continuously tracked by charge nurse). Patients who are medically ready for transfer out have an accepting service in place and a bed ready on the floor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in alarm rate before and after intervention | 24 hours before intervention and 72 hours after intervention
  Within-subject comparison evaluating the numbers of alarms and the trajectories of alarm rates in the 24 hours before and up to 72 hours after each huddle

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Bonafide, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States